CLINICAL TRIAL: NCT04466631
Title: SAlute e LaVoro in Chirurgia Oncologica (SALVO)
Brief Title: Health and Employment After Gastro Intestinal Surgery - HEAGIS2
Acronym: HEAGIS2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Collaborators: Humanitas Hospital, Italy (Other); Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 232050b
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-06

CONDITIONS: Esophageal Neoplasms; Gastric Neoplasm; Colon Neoplasms
Keywords: quality of life; employment; social activities; surgery
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observative longitudinal: The participants won't receive any support during the post surgery period.

SUMMARY:
By using the M.A.D.I.T. methodology and the Dialogics science, SALVO Project aims to develop operational guidelines to support oncological target patients in the resumption of their daily post-operative activities. The research will implement an instrument for the purpose of measuring the health need of participants who are admitted to the surgical ward. Therefore, targeted interventions will be implemented with participants, and efficacy will be evaluated in order to define treatment guidelines.

The principal aim of this study is to create a validated and replicable intervention model for supporting patients who undergone surgery for esophageal and gastro intestinal cancer.

DETAILED DESCRIPTION:
Several studies highlight how patients diagnosed with a digestive tract cancer, experience difficulties in returning to work after treatment, leading to socio-economic spill-over effects.

A specific 16 questions questionnaire had been developed for this study, the "Health and Employment After Gastro Intestinal Surgery Dialogical Questionnaire" (HEADS-DQ). It investigate peculiar patient competences involved after surgery: future forethought; context evaluation; consequences of own actions forethought; use of available resources, each relevant to four areas: clinical; familiar; working; daily-activities.

Through this questionnaire participants ability in dealing with after surgery consequences will be evaluated in order to describe their development during the post surgery period.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old;
* Comprehension of Italian language;
* Esophageal or gastrointestinal cancer diagnosis;
* Curative surgery;
* No metastasis or neoplasm recurrence.

Exclusion Criteria:

* <18 years old;
* No comprehension of Italian language;
* Not esophageal or gastrointestinal cancer diagnosis;
* Palliative surgery;
* Metastasis or neoplasm recurrence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergone surgery for esophagus or gastrointestinal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Utilization of specific competences by participants | 9 months after the surgery
  Textual data derived from textual analysis: future forethought; context evaluation; consequences of own actions forethought; use of available resources, each relevant to four areas: clinical; familiar; working; daily-activities

SECONDARY OUTCOMES:
Number of participants maintaining their job | 9 months after the surgery
Number of participants with jejunostomy maintaining their job | 9 months after the surgery
Number of participants maintaining their social activities | 9 months after the surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Humanitas Mirasole S.p.a., Rozzano, Milan
  - Istituto Oncologico Veneto - IOV IRCSS, Castelfranco Veneto, Treviso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Blasi G, Bouteyre E, Rollin L. Giving up work after cancer: An exploratory qualitative study of three clinical cases. Work. 2018;60(1):105-115. doi: 10.3233/WOR-182712. PMID 29733033
- [Background] Moran JR, Short PF, Hollenbeak CS. Long-term employment effects of surviving cancer. J Health Econ. 2011 May;30(3):505-14. doi: 10.1016/j.jhealeco.2011.02.001. Epub 2011 Mar 1. PMID 21429606
- [Background] Yarker J, Munir F, Bains M, Kalawsky K, Haslam C. The role of communication and support in return to work following cancer-related absence. Psychooncology. 2010 Oct;19(10):1078-85. doi: 10.1002/pon.1662. PMID 20014202
- [Background] Parsons JA, Eakin JM, Bell RS, Franche RL, Davis AM. "So, are you back to work yet?" Re-conceptualizing 'work' and 'return to work' in the context of primary bone cancer. Soc Sci Med. 2008 Dec;67(11):1826-36. doi: 10.1016/j.socscimed.2008.09.011. Epub 2008 Oct 11. PMID 18851893
- [Background] Mehnert A. Employment and work-related issues in cancer survivors. Crit Rev Oncol Hematol. 2011 Feb;77(2):109-30. doi: 10.1016/j.critrevonc.2010.01.004. Epub 2010 Feb 8. PMID 20117019
- [Background] Pinto E, Cavallin F, Alfieri R, Saadeh LM, Mantoan S, Cagol M, Castoro C, Scarpa M. Impact of esophagectomy for cancer on patients' occupational status. Eur J Surg Oncol. 2016 Jan;42(1):103-9. doi: 10.1016/j.ejso.2015.09.021. Epub 2015 Oct 9. PMID 26482347
- [Background] Martinez LR, White CD, Shapiro JR, Hebl MR. Selection BIAS: Stereotypes and discrimination related to having a history of cancer. J Appl Psychol. 2016 Jan;101(1):122-8. doi: 10.1037/apl0000036. Epub 2015 Jun 29. PMID 26121089
- [Background] Clarke TC, Christ SL, Soler-Vila H, Lee DJ, Arheart KL, Prado G, Caban-Martinez A, Fleming LE. Working with cancer: health and employment among cancer survivors. Ann Epidemiol. 2015 Nov;25(11):832-8. doi: 10.1016/j.annepidem.2015.07.011. Epub 2015 Aug 4. PMID 26320705
- [Background] Turchi GP, Iudici A, Faccio E. From Suicide Due to an Economic-Financial Crisis to the Management of Entrepreneurial Health: Elements of a Biographical Change Management Service and Clinical Implications. Front Psychol. 2019 Mar 4;10:426. doi: 10.3389/fpsyg.2019.00426. eCollection 2019. No abstract available. PMID 30886599
- [Background] Iudici A, Favaretto G, Turchi GP. Community perspective: How volunteers, professionals, families and the general population construct disability: Social, clinical and health implications. Disabil Health J. 2019 Apr;12(2):171-179. doi: 10.1016/j.dhjo.2018.11.014. Epub 2018 Nov 29. PMID 30528178